CLINICAL TRIAL: NCT05086705
Title: Cool Down With EMBr: Enhancing Menopausal Hot Flash Symptom Reduction After Breast Cancer
Brief Title: EMBr Wave for the Reduction of Hot Flashes in Women With a History of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Embr Labs, Inc. (Industry)
Responsible Party: Principal Investigator, Sagar Sardesai, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-19152; NCI-2019-05843 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Carcinoma; Breast Ductal Carcinoma In Situ; Breast Lobular Carcinoma In Situ; Hot Flashes
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A (EMBr Wave) (Experimental): Patients utilize the EMBr Wave device for 4 weeks, then crossover to arm B for 4 weeks.
  Interventions: Device: EMBr Wave; Other: Questionnaire Administration
- Arm B (crossover) (Active Comparator): Patients receive no treatment for 4 weeks, then crossover to arm A for 4 weeks.
  Interventions: Device: EMBr Wave; Other: Questionnaire Administration

INTERVENTIONS:
Device: EMBr Wave — Use EMBr Wave
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well EMBr Wave technology works in reducing hot flashes in women with a history of breast cancer. Hot flashes are a common symptom experienced by menopausal women. The standard treatment for hot flashes is hormone replacement therapy, however hormone replacement therapy cannot be used in women with a history of, or active, breast cancer. EMBr Wave is a personal heating and cooling device worn on the wrist. EMBr Wave may help reduce hot flash severity in women with a history of breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of using EMBr Wave technology in women with a history of breast cancer who are experiencing bothersome hot flashes.

SECONDARY OBJECTIVES:

I. To evaluate the preliminary efficacy of EMBr Wave in reducing hot flash severity and frequency in women with a history of breast cancer.

II. To identify in what ways EMBr Wave has the greatest potential efficacy, such as reduction in vasomotor symptoms (VMS) severity, frequency, duration, sense of control, or self-esteem.

III. To estimate effect sizes to inform power calculations for a future phase III trial.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients utilize the EMBr Wave device for 4 weeks, then crossover to arm B for 4 weeks.

ARM B: Patients receive no treatment for 4 weeks, then crossover to arm A for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with history of breast cancer, ductal breast carcinoma in situ (DCIS), or lobular breast carcinoma in situ (LCIS) (currently without evidence of malignant disease)
* Bothersome hot flashes (defined by their occurrence of >= 28 times per week and of sufficient severity to prompt the patient to seek therapeutic intervention)
* Presence of hot flashes for > 30 days prior to study entry
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to wear EMBr Wave device during the study period
* Willingness to use the EMBr Wave mobile application
* Have a working smartphone that can download the EMBr Wave mobile application (iPhone 6 or more recent generation, Android 8.0 or more recent generation)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) = 0, 1
* Ability to provide informed written consent
* Life expectancy >= 6 months

Exclusion Criteria:

* Antineoplastic chemotherapy (anti-HER2 agents allowed) (current [=< 4 weeks prior] or planned therapy)
* Androgens (current [=< 4 weeks prior] or planned therapy)
* Systemic estrogens. Local vaginal estrogen preparations are allowed, but need to have been initiated for vulvo-vaginal atrophy at least 28 days prior, and must not be expected to stop or change the dose or frequency of the medication during the study period (current [=< 4 weeks prior] or planned therapy)
* Progestogens (current [=< 4 weeks prior] or planned therapy)
* Tamoxifen, raloxifene and aromatase inhibitors are allowed, but patient must have been on a constant dose for at least 28 days and must not be expected to stop the medication during the study period (current [=< 4 weeks prior] or planned therapy)
* Selective serotonin reuptate inhibitors (SSRIs)/serotonin-norepinephrine reuptake inhibitor (SNRIs), when being used for hot flash management or other indications such as depression, is allowed, assuming the dose will remain unchanged for the study duration (current [=< 4 weeks prior] or planned therapy)
* Gabapentin/pregabalin, when being used for hot flash management (use for other indications, such as pain, is allowed, assuming the dose will remain unchanged for the study duration) (current [=< 4 weeks prior] or planned therapy)
* Clonidine (current [=< 4 weeks prior] or planned therapy)
* Prior use of EMBr Wave
* Nickel allergy
* Pregnant or nursing women since the safety of device has not been established in this population

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Sardesai, MBBS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (EMBr Wave First): Patients utilize the EMBr Wave device for 4 weeks, then receive no treatment for 4 weeks.
  EMBr Wave: Use EMBr Wave
  Questionnaire Administration: Ancillary studies
- Arm B (EMBr Wave Second): Patients receive no treatment for 4 weeks, then utilize the EMBr Wave Device for 4 weeks.
  EMBr Wave: Use EMBr Wave
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm A (EMBr Wave First) | Arm B (EMBr Wave Second)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (EMBr Wave First) | Arm B (EMBr Wave Second) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 48
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Device Usage
Description: Feasibility will be evaluated primarily with respect to device usage. The proportion of patients who wear the device for at least 8 hours between 8:00 am and 8:00 pm for at least 22 days will be estimated using the entire sample and a 95% Jeffreys interval for binomial proportions will be computed.
Time Frame: Up to 8 weeks
Population: Data was not collected or analyzed
Arm/Group | Arm A (EMBr Wave First) | Arm B (EMBr Wave Second)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Patient Satisfaction
Description: Feasibility will be evaluated secondarily with respect to patient satisfaction. The mean patient satisfaction scores for each Likert-type question and proportion of patients reporting satisfaction scores at or above 7 will be estimated in the entire sample and compared between sequence groups at the 5% significance level (two-sided).Rated on a 10-point Likert scale with 10 being most satisfied or most effective.
Time Frame: At 8 weeks
Population: Patient satisfaction data was only obtained for the 29 out of 50 participants who gave responses for the exit survey (12 from Arm A and 17 from Arm B). Satisfaction scores pertain to satisfaction with EMBr wave device usage, so no data is reported for the No Treatment Group
Measure: Mean (Full Range); unit: score on a scale
Groups:
- EMBr Wave Device: Patients utilize the EMBr Wave device for 4 weeks.
- No Treatment: Patients receive no treatment for 4 weeks.
Arm/Group | EMBr Wave Device | No Treatment
Number analyzed (Participants) | 29 | 0
score on a scale
  Intensity | 4.97 [0 to 10] |
  Duration | 5.48 [0 to 10] |
  Work | 4.76 [0 to 10] |
  Social | 4.72 [0 to 10] |
  Leisure | 4.86 [0 to 10] |
  Sleep | 4.41 [0 to 10] |
  Mood | 4.97 [0 to 10] |
  Concentrate | 4.90 [0 to 10] |
  Relation | 4.41 [0 to 10] |
  Sexuality | 3.24 [0 to 10] |
  Enjoy | 5.10 [0 to 10] |
  Quality | 5.38 [0 to 10] |
  Worth | 5.79 [0 to 10] |
  Satisfy | 5.52 [0 to 10] |

3. Secondary Outcome: Effect of EMBr Wave Using Hot Flash-Related Daily Interference Scale (HFRDIS)
Description: Reported via patient reported outcomes, primarily Hot Flash-Related Daily Interference Scale (HFRDIS), a scale of 0-10 with 0 being no interference (best outcome) and 10 being completely interfere (worst outcome). Survey administered on paper or via RedCap survey distribution at week 4 and week 8.
Time Frame: At week 4 and at week 8
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- EMBr Wave Device: Participants utilized the EMBr wave device for 4 weeks.
- No Treatment: Patients received no treatment for 4 weeks.
Arm/Group | EMBr Wave Device | No Treatment
Number analyzed (Participants) | 50 | 50
units on a scale
  Work | 3.6368 (0.3386) | 3.6743 (0.3261)
  Social Activities | 3.0626 (0.3356) | 3.1652 (0.3590)
  Leisure Activities | 3.4362 (0.3063) | 3.5256 (0.3566)
  Sleep | 4.8231 (0.3948) | 5.4950 (0.3403)
  Mood | 3.7743 (0.3367) | 4.0794 (0.3254)
  Concentration | 3.7391 (0.3464) | 4.1341 (0.3634)
  Relations with others | 2.5774 (0.3331) | 2.6717 (0.3520)
  Sexuality | 2.9739 (0.4058) | 3.1144 (0.4228)
  Enjoyment of Life | 3.2259 (0.3234) | 3.3231 (0.3651)
  Quality of Life | 3.4489 (0.3248) | 3.5543 (0.3386)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the study duration; a total 8 months.
Arm/Group | EMBr Wave Device | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT05086705/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT05086705/ICF_001.pdf